CLINICAL TRIAL: NCT06987552
Title: A Pilot Study of Single-Port Robot-Assisted Surgery Using Da Vinci SP Surgical System for Patients With Upper Tract Urothelial Cancer
Brief Title: Single-Port RAS Using Da Vinci SP Surgical System for UTUC Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202409016DIPD
Record Dates: First submitted 2025-02-25; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-12

CONDITIONS: Upper Tract Urothelial Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Operation of focus procedure with da Vinci SP Surgery System (Experimental): Single-Port Robot-Assisted Surgery Using Da Vinci SP Surgical System for Patients with Upper Tract Urothelial Cancer
  Interventions: Device: Da Vinci SP Surgical System

INTERVENTIONS:
Device: Da Vinci SP Surgical System — Da Vinci SP Surgical System

SUMMARY:
To evaluate patient-reported outcomes of radical nephroureterectomy using single-port robotic surgery

DETAILED DESCRIPTION:
To evaluate safety, surgical outcomes, patient characteristics, and patient-reported outcomes of radical nephroureterectomy using single-port robotic surgery

ELIGIBILITY:
Inclusion Criteria:

* Age 20 years or more
* Histologically or cytologically diagnosed upper tract urothelial cancer
* Fitting indications of radical nephroureterectomy and ipsilateral bladder cuff resection, and deemed feasible for robotic surgery
* ASA physical status classification 1-2 and adequate organ function
* Patients willing and able to comply with study protocol requirements and follow-up
* With informed consent

Exclusion Criteria:

* Synchronous bladder cancer
* Distant metastasis of cancer
* BMI ≥30 or BMI <18.5
* Unable to tolerate lateral decubitus or Trendelenburg position (relative contra-indication)
* Severe adhesion due to prior abdominopelvic surgery (relative contra-indication)
* Previous radiation treatment to the pelvic area
* Active infectious disease
* Severe concomitant illness that drastically shortens life expectancy or increases risk of therapeutic interventions, such as: severe heart disease (NYHA functional class III-IV) or severe lung disease (GOLD Group C-D)
* Cannot follow trial-required procedures
* Concomitant systemic or pelvic disease that increases the risk of surgery
* Long-term use of anti-coagulant(s)
* Patients with coagulopathy
* Emergency surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of conversion rate | During Surgery
  The primary performance endpoint will be assessed as the ability to successfully completed the planned procedure with da Vinci SP System, with no conversion to alternative surgery including open surgery or laparoscopy.

SECONDARY OUTCOMES:
Perioperative Parameters: Operative Time | immediately after the surgery
  First skin incision to closure of wound by minutes.
Perioperative Parameters: Console Time | immediately after the surgery
  Surgeon on Console Time by minutes
Perioperative Parameters: Transfusion | immediately after the surgery
  Blood transfusion amount by bags
Perioperative Parameters: Estimated Blood Loss | immediately after the surgery
  Estimated blood loss by mL
Postoperative Parameters: Length of Stay | 30 days post operation
  Total length of stay = discharge date - admission date
Complication | 30 days post operation
  Intraoperative and/or postoperative complication rate in 30 days by Clavien-Dindo Classification
Postoperative Parameters: Readmission | 30 days post operation
  Readmission rate by %
Postoperative Parameters: Reoperation | 30 days post operation
  Reoperation rate by %
Perioperative Mortality | 30 days post operation
  Mortality by %
Pain Score | 30 days post operation
  measured by Visual Analogue Scale (VAS) for pain assessment at baseline, post operation, and discharge day. VAS ranged from 0 to 10, representing no pain to extreme pain.

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Chieh Chueh, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/52/NCT06987552/Prot_000.pdf